CLINICAL TRIAL: NCT02382354
Title: Comparison of the Effect-site Concentration of Remifentanil for Insertion of the I-gel and Laryngeal Mask Airway During Propofol Anesthesia
Brief Title: Remifentanil for the I-gel and Laryngeal Mask Airway Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-14-417
Record Dates: First submitted 2015-02-25; First posted 2015-03-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Supraglottic Airways for General Anesthesia
MeSH Terms: interventions — Remifentanil; Laryngeal Masks; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- i-gel (Experimental): I-gel insertion was attempted during propofol and remifentanil anesthesia .
  Interventions: Drug: remifentanil; Device: i-gel; Drug: propofol
- laryngeal mask airway (Active Comparator): LMA insertion was attempted during propofol and remifentanil anesthesia .
  Interventions: Drug: remifentanil; Device: laryngeal mask airway; Drug: propofol

INTERVENTIONS:
Drug: remifentanil — The predetermined effect-site concentration of remifentanil was started using modified Dixon's up-and-down method
  Other Names: ultiva
Device: i-gel — I-gel insertion was inserted 5 min after anesthesia induction
  Arms: i-gel
Device: laryngeal mask airway — laryngeal mask airway insertion was inserted 5 min after anesthesia induction
  Arms: laryngeal mask airway
Drug: propofol — Anesthesia was induced with propofol target-controlled infusion at the effect-site concentration of 5 μg/ml
  Other Names: fresofol

SUMMARY:
Structural differences of supraglottic airway devices could influence the different compressive forces in the oropharyngeal cavities, and require different depth of anesthesia. The addition of remifentanil during propofol anesthesia facilitates the insertion of laryngeal mask airway (LMA) with minimal adverse hemodynamic disturbances. This study was designed to determine the effect-site concentration of remifentanil in 50% of patients (EC50) and 95% of patients (EC95) for successful i- gel insertion, and compare those for LMA insertion during propofol target-controlled infusion (TCI).

DETAILED DESCRIPTION:
Anesthesia was induced with propofol TCI at the effect-site concentration of 5 μg/ml, and the predetermined effect-site concentration of remifentanil was started simultaneously. The remifentanil concentration was determined using modified Dixon's up-and-down method (initial concentration: 3.0 ng/ml, step size: 0.5 ng/ml). Five minutes later, i- gel or LMA insertion was attempted. The response of the patients to the insertion of LMA was classified as either 'movement' or 'no movement'.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing general anesthesia for short elective surgery (<2 hr)

Exclusion Criteria:

* G-E reflux
* obesity (BMI>30)
* anticipated difficult airway

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
successful insertion of i-gel and LMA | from 5 min after anesthetic induction to 1min after device insertion

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University hospital, Suwon, South Korea